CLINICAL TRIAL: NCT03395925
Title: Evaluation of the Thyroid Volume After Radiofrequency Ablation of Thyroid Nodules and Recurrent Thyroid
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not started
Sponsor: Olympus Surgical Technologies Europe (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEL THYRO01
Record Dates: First submitted 2017-12-17; First posted 2018-01-10 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Thyroid Nodule
Keywords: Thyroid Nodule; Bipolar coagulation electrode; radiofrequency ablation
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Celon Pro Surge (Experimental): Ablation of thyroid tissue
  Interventions: Device: Celon Pro Surge

INTERVENTIONS:
Device: Celon Pro Surge — bipolar coagulation electrode intended for tissue heating
  Other Names: Bipolar coagulation electrode, tissue heating and ablation

SUMMARY:
Thyroid nodules are among the common alterations of the thyroid. Depending on the detection method the prevalence is between 20% and 50%, whereas the incidence increases with improvement of ultrasonic technology. The CelonPro Surge bipolar coagulation electrode operated with the compatible power control unit and compatible tube pump is indicated for ablation and coagulation of soft tissue, including thermal inactivation and/or volume reduction of locally defined tissue areas, such as tumors and metastases.

The primary objective of the study is to assess the influence of radiofrequency ablation due to thyroid volume after 24 hours, 3 months, 6 months and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given written (personally signed and dated) informed consent before completing any study-related procedures (i.e. any assessment or evaluation that would not have formed part of their normal medical care).
* The patient must be aged 18yrs or older.
* The patient must be able to understand, and be willing to comply with the requirements of the protocol
* The patient is not pregnant
* The patient has the diagnosis of benign thyroid nodules, struma diffusa, struma uninodosa, struma multinodosa, struma per magna, Thyroidea nodosa or Thyroidea multinodosa
* The patient rejected surgery The patient rejected sole radioiodine therapy

Exclusion Criteria:

* Malign nodules
* Pregnancy
* Pacemaker near the target issue (<4cm)
* Nerve stimulating device
* High fever
* Prosthesis for the inner ear

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
The primary objective of the study is to demonstrate reduction of thyroid volume following radiofrequency ablation of thyroid tissue | 1 year
  The primary endpoint is the reduction of thyroid volume at 12-Month follow-up visit. A responder to the radiofrequency treatment is defined as a subject with any reduction of the thyroid volume.

CONTACTS AND LOCATIONS:
Overall Officials: Hüdayi Korkusuz, Prof., Principal Investigator — Goethe University
Locations (1):
- Johann-Wolfgang Goethe University, Frankfurt, Germany

IPD SHARING:
Plan to Share IPD: No